CLINICAL TRIAL: NCT05015881
Title: Relationship Between Brain and Heart Glucose Metabolism in Alcohol Use Disorder
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 848992
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder (AUD); Alcohol Drinking
Keywords: Ester Keytone; MRI; PET scan; Echocardiogram
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — rVSV-deltaG-spike COVID-19 vaccine; Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Randomized, 2-way crossover trial in 10 individuals with AUD and 10 Healthy controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketone ester + echocardiogram + PET FDG scanning visit. (Active Comparator): Subjects will drink single dose of ketone ester 1.9 kcal/kg + echocardiogram + PET scanning visit. Dietary Supplement: Ketone Ester "(R)-3-hydroxybutyl (R)-3-hydroxybutyrate" (R)-3-hydroxybutyrate (commercially available as DeltaG, (TdeltaS, Orlando, FL). 2-Deoxy-2-[18F] fluoro-D-glucose (FDG) Positron Emission Tomography/Computed Tomography (PET/CT) scan.
  Interventions: Dietary Supplement: Ketone Ester "(R)-3-hydroxybutyl (R)-3-hydroxybutyrate"; Drug: FDG
- Echocardiogram + PET FDG scanning visit. (Other): Subjects will complete a echocardiogram + PET scanning visit. 2-Deoxy-2-[18F] fluoro-D-glucose (FDG) Positron Emission Tomography/Computed Tomography (PET/CT) scan.
  Interventions: Drug: FDG

INTERVENTIONS:
Dietary Supplement: Ketone Ester "(R)-3-hydroxybutyl (R)-3-hydroxybutyrate" — Drink a single dose of ketone ester 1.9 kcal/kg
  Other Names: DeltaG
  Arms: Ketone ester + echocardiogram + PET FDG scanning visit.
Drug: FDG — Echocardiogram, and 2-Deoxy-2-[18F] fluoro-D-glucose (FDG) PET scan.
  Other Names: 2-Deoxy-2-[18F] fluoro-D-glucose (FDG)

SUMMARY:
The goal of this study is to learn more about how a nutritional supplement "ketone ester" (deltaG ®) has an effect on brain and heart function and on alcohol consumption in individuals with and without alcohol use disorder. The study will use Fluorodeoxyglucose (FDG) Positron Emission Tomography/Computed Tomography (PET/CT) scans after a single dose of ketone ester or Placebo in 10 people with alcohol use disorder and 10 healthy control volunteers.

DETAILED DESCRIPTION:
The purpose of this research is to study how a nutritional ketone ester may affect brain and heart function in individuals who consume alcohol on a regular basis, and in healthy controls.

The study will see how the brain and heart responds, once after drinking the ketone ester and once without drinking the ester (baseline) using a test called an FDG PET/CT scan. PET/CT scans use small amounts of a radioactive imaging drug, a special camera and a computer to evaluate organ and tissue functions. FDG PET/CT scans are routinely done for evaluation of heart diseases. The study will test how the brain and heart function at rest and while viewing pictures of alcohol.

The study involves 4 or more visits: (1) a consent/screening visit, which can be completed in a single day or divided over multiple days. Portions of the screening may occur using telephone or video conference. (2) In-person MRI (if one hasn't been completed in the past year). (3) In-person study visit that includes the drinking of the ketone ester, a FDG PET/CT scan, and (4) a second in-person visit that a FDG PET/CT scan without drinking the ketone ester. Depending on the scheduling for each of these visits, study involvement will last approximately 8 weeks depending on scheduling restrictions. Following completion of the scan visits (next business day), study staff will follow-up with individuals by phone to ask about any changes to your health and to ensure that they did not experience any side effects from the ketone ester, MRI scan or FDG PET/CT scan.

Screening visit:

* Informed consent will happen before any study related procedures are performed. Staff will answer all questions during the process. The following will occur at the screening session:
* Demographic information, such as date of birth, age, biological sex, race, and ethnicity will be collected.
* Current address and contact information in order to register people into the University of Pennsylvania electronic medical record system.
* Collection of a urine sample of about 30 mL (approximately 2 tablespoons) to be used for urinalysis, drug screening and pregnancy in women.
* Breathalyzer test to measure breath alcohol concentration (BrAC). A 0.000% BrAC is required to continue with the visit.
* Vitals (blood pressure and pulse), weight and height. A doctor or nurse practitioner will do a brief physical exam.
* Brief psychiatric assessments called the 'CSSRS'. During these interviews, questions will be asked about current and past depressed mood symptoms, as well as other psychiatric symptoms, including suicidal thinking.
* Complete a brief mental ability test called the 'Shipley Institute of Living Scale'.
* Short interview regarding alcohol and smoking history, behaviors, and mood and any drug or alcohol use, and questions about any substance cravings or withdrawal symptoms.
* Psychological questionnaires related to substance use, cravings, risk behaviors, mental health, personality, depression and anxiety, quality of sleep.
* Complete questions about any current medication, recreational drugs or supplements use.
* Complete a questionnaire about the presence of metal in the body to determine if it is safe to undergo an MRI.
* A small amount of blood (approximately 2.75 tablespoons) will be drawn for screening lab tests (a blood count and chemistry panel), genetics and metabolite analysis.
* Complete an oral swab rapid HIV test. If the test is positive, study staff will draw a tablespoon of blood to conduct a confirmatory HIV blood test (i.e., to confirm the positive oral test). If the blood test are positive for HIV, we will provide a referral for medical care and a copy of the test results.
* Complete several computer-based tasks on a laptop that will be provided by the study team. These tasks will test the following brain cognition measures including: visual memory, willingness to delay a reward offered, response time in reacting to specific information on the screen, verbal learning and memory, impulsiveness, and reaction time and accuracy when asked to match up a series of test pictures that are different shapes and colors.

Results of the screening visit, will be available within 2 weeks to confirm if eligibility to continue with the study and schedule the rest of the study visits.

A Brain MRI scan visit (1 hour):

Scheduled if there was not an MRI in the past year. An MRI is a test that uses a magnetic field and pulses of radio wave energy (pulse sequences) to make pictures of your brain. A small meal will be provided before the MRI. MRI images are collected in a Magnetic Resonance Imaging scanner. The MRI scan will be done to understand brain anatomy (the structure of the brain) and the function of the brain during rest and when looking at pictures of alcohol. The MRI will last up to 1 hour.

* Complete a MRI safety form
* Remove any metal from the body
* Earplugs are provided for the noise from the MRI scanner, and subjects will be positioned on the imaging table with head in the scanner, held comfortably in a special head holder.
* Undergo several scans (up to 60 minutes in total). Subjects will be instructed not to move the head and to lie as still as possible during the scan (up to 60 minutes).
* Complete a Cue Reactivity task during the scan. In this task involves viewing pictures of various items such as food or alcohol on the screen. Subjects will rate the items by pressing a button. The task will take up to 10 minutes to complete.

PET Scanner Visits (this will last 3-4 hrs):

Subjects are asked to fast for 6 hours prior to the PET scanning visits. On the day of the study visits the following will be done:

* Meet a study team member at the Hospital of the University of Pennsylvania.
* Take a Breathalyzer test to measure breath alcohol concentration. Must have a 0.000% BrAC to continue with the visit.
* Complete questions about recent use drugs, alcohol, nicotine, and substance use and then asked to give a urine sample. This will be used for a rapid urine drug test. Positive test will be reviewed by the study doctor to determine if visit may continue. Woman of childbearing potential will receive a urine pregnancy test. The result of the pregnancy test must be negative to continue to participate in the study.
* Trained staff will placed two IVs to draw blood and give the FGD tracer. Staff will measure vitals (blood pressure and pulse), weight and height.
* A list of current medications and vitamins will be reviewed to determine any changes in medications, dosage or frequency of use of any medications or vitamins since the screening visit.
* A ketone ester drink will be given on one of the 2 scan visits. There will be two study visits that have the same procedures, except that on one study day subjects are asked to drink a drink with the ketone ester, and on the other visit not drink the ketone ester.
* Staff will perform an Echocardiography. This is an ultrasound of the heart.
* Once the Echocardiography is complete, subjects will undergo a Positron Emission Tomography / Computed Tomography (PET/CT) with FDG scan for approximately 60 minutes
* Imaging of FDG is done with specialized cameras that can pick up the tiny radiation signals given off by the radiotracer and determine where the signals come from. In this way, we can form a picture of where the radiotracer goes after it is injected. The type of scan is called a PET/CT scan, which uses a large doughnut shaped detection device to provide a map of where radiotracers go in the body.
* Subject will be asked to remove any metal objects before entering the scanner. The FDG tracer will be injected using the IV after positioning on the scanner. Subjects will lie face up on the scanner table for about 1 hour, while the PET/CT machine collects imaging information over the body. Blood samples will be drawn before the injection and at 5 other time points during the scan. Approximately 45 mL (about 9 teaspoons) of blood will be collected during the scan. The blood will be used to measure radioactive counts and/or test how the tracer is being metabolized by the body.

Follow-up Staff will call to ask about any uncomfortable symptoms at any time during the imaging scan process or in the 24 hours (day or night) following the study visits.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for both study groups (AUD and controls)

  1. Age 21 years to 65 years old.
  2. Willingness to provide signed, informed consent and commit to completing the procedures in the study
  3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.
  4. Participants must agree to not consume alcohol beverages for 24 hours prior to each laboratory session.

     Inclusion criteria for the AUD group:
  5. Meets DSM-5 criteria for current AUD
  6. Participants report average weekly ethanol consumption of at least 15 standard drinks weekly over the past month prior to consent (self-report)
  7. Minimum 1 year history of heavy drinking (self-report).
  8. Must have had last drink within 1 week of PET visits.
  9. Alcohol specified as the preferred drug (self-report).

     Inclusion criteria for the control group:
  10. AUDIT score < 6
  11. Drinks alcohol 15 standard drinks or less per month and 3 or less standard drinks per occasion.

Exclusion both groups:

1. Females who are pregnant or breast-feeding will not be eligible for this study. Female participants of child-bearing potential will have a urine pregnancy test prior to FDG injection.
2. Unwilling or unable to refrain from use, within 24 hours of FDG PET/CT scan procedures, psychoactive medications or medication that may affect study results (e.g., analgesics containing narcotics, antibiotics, anti-inflammatory drugs).
3. Current DSM-5 diagnosis of a major psychiatric disorder (other than nicotine use disorders, or marijuana use disorders that are mild/moderate in both groups; and alcohol in the AUD group) that required hospitalization, or that required daily medications for over 4 weeks in the past year (i.e., antidepressants; anticholinergics; antipsychotics; anxiolytics; lithium; psychotropic drugs not otherwise specified (nos) including herbal products (no drugs with psychomotor effects or with anxiolytics, stimulant, antipsychotic, or sedative properties); sedatives/hypnotics).
4. Positive urine drug screen positive for any substances, other than marijuana, on study visits (may be repeated once and if the result is negative on repeat it is not exclusionary).
5. Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.
6. Currently suffering from or with a history of stroke and/or stroke related spasticity per medical record review or self report.
7. History of seizures per medical record review or self report.
8. HIV positive, as the human immunodeficiency virus may affect the brain, per medical record review or self report or by testing at screening.
9. Head trauma with loss of consciousness for more than 30 minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI. (self-report, medical record review).
10. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head, fear of enclosed spaces, or other standard contraindication to MRI (self-report checklist) or PET scanner.
11. Significant claustrophobia or other medical condition preventing subject from lying comfortably flat on his/her back for up to 2 hours in the MRI or PET scanner (self-report).
12. BMI > 35, imaging data acquisition is impaired with high-weight individuals).
13. Vision problems that cannot be corrected with glasses.
14. Judged by the principal investigator or his designee to be an unsuitable candidate for study participation.

    Exclusion criteria for the control group:
15. Current DSM-5 diagnosis of Alcohol use disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
FDG uptake (CMRg) in the brain and heart | 4 hours
  The primary outcome measure to be analyzed is a comparisons of AUD subjects and healthy control subjects in the amount of FDG uptake (CMRg metabolic rate of glucose) in brain and heart.

SECONDARY OUTCOMES:
Amount of FDG uptake (CMRg) | 4 hours
  The secondary outcome measure is the comparisons of ketone ester intervention versus intervention in FDG uptake (CMRg metabolic rate of glucose) in AUD subjects versus health control subjects.
Amount of blood glucose (mmol/L or mg/dl) | 4 hours
  Third outcome measure is the comparisons of ketone ester intervention versus intervention in blood glucose levels in AUD subjects versus health control subjects.
Amount of BHB (beta-hydroxybutyrate) (mmol/L) | 4 hours
  Fourth outcome measure is the comparisons of ketone ester intervention versus intervention in BHB (beta-hydroxybutyrate) (mmol/L) levels in AUD subjects versus health control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde E Wiers, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States